CLINICAL TRIAL: NCT03790436
Title: A Pilot Study on the Feasibility and Tolerability of Betaquik, a Special Medical Food Containing Medium Chain Triglycerides (MCT) as an Adjunct to the Dietary Management of Epilepsy and Quality of Life in Adults on the Modified Atkins Diet (MAD)
Brief Title: Betaquik as an Adjunct to Dietary Management of Epilepsy in Adults on the Modified Atkins Diet
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We no longer have Ketogenic Dietician coverage/access.
Sponsor: University of Southern California (Other)
Collaborators: Vitaflo International, Ltd (Industry)
Responsible Party: Principal Investigator, Arthur Partikian, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-17-01011
Record Dates: First submitted 2018-11-20; First posted 2018-12-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Epilepsy; Epilepsy Intractable; Seizures; Seizure Disorder; Ketogenic Dieting; Ketosis
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy; Seizures; Ketosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Betaquik (Experimental)
  Interventions: Dietary Supplement: Betaquik

INTERVENTIONS:
Dietary Supplement: Betaquik — Study dietitian will advise each participant on target volume of Betaquik (45g MCT, 225mL Betaquik). Consuming too much MCT too quickly may cause gastrointestinal discomfort such as abdominal pain or diarrhea, this is related to its assimilation to the body. Any symptoms that do occur normally resolve in the majority of patients, and with time and persistence, GI tolerance is usually established.
  Therefore the study dietitian will advise on a gradual systematic introduction to minimize any adverse effects. The daily-tolerated amount will be divided into 3-4 equal portions, taken regularly throughout the day. subjects will be advised to always take Betaquik with food, as part of meals and snacks, to help promote gastrointestinal tolerance. The goal is within the first 4 weeks participants will have reached their tolerated target volume of Betaquik.

SUMMARY:
The purpose of this pilot study is to measure adherence and quality of life in adults with intractable epilepsy following the Modified Atkins Diet (MAD) with Betaquik, a ready-to-use medium chain triglyceride (MCT) emulsion, as an adjunct to the MAD.

DETAILED DESCRIPTION:
The purpose of this pilot study is to measure adherence and quality of life in adults with intractable epilepsy following the Modified Atkins Diet (MAD) with Betaquik, a ready-to-use medium chain triglyceride (MCT) emulsion, as an adjunct to the MAD.

The participants dietitian will recommend an appropriate daily intake of Betaquik based on individual requirements. Participants will be asked to gradually introduce Betaquik into the diet up to the target volume advised by the dietitian. Participants will then incorporate the target volume of Betaquik into their diet and gradually increase carbohydrate intake up to a maximum tolerated level and continue on the management regime until the end of the 26-week period. At the end of the 26-week period participants will undergo a Betaquik washout. In order to mitigate any impact of Betaquik tapering dietary effectiveness and sustained ketosis, carbohydrate intake will be reduced concurrently to the original 20-30 grams daily. This will continue for an additional 26-weeks (totaling 52-weeks). Both Betaquik introduction and tapers will occur under the direction of their dietitian with their daily intake under weekly review for the duration of the study. Vitaflo International Ltd. will supply Betaquik directly to the participants homes free of charge. Participants will be provided with a 28-day supply of Betaquik renewed every four weeks.

The objective of this study is to evaluate the acceptability, tolerance and adherence of the MAD including MCT - Betaquik in participants with a diagnosis of epilepsy.

This is an exploratory pilot study to evaluate the gastrointestinal tolerance, palatability and participant adherence, over a 52-week period, of the MAD with and without Betaquik, for the dietary management of participants with epilepsy.

Participants will be asked to collect daily information on any incidence of the following for the first 3 months and weekly thereafter:

* Diarrhea and/or constipation as measured by stool frequency, color and consistency
* Bloating and/or distension
* Nausea and/or vomiting
* Burping/flatulence/regurgitation
* Abdominal discomfort/pain

If participants report any of the above then additional questions about the timing, duration, cause and seriousness/severity of any adverse effects are to be recorded in the diary.

At the end of the 52-weeks all final questionnaires will be completed including those assessing quality of life, clinical epilepsy status, dietary intake and adherence, Betaquik and dietary carbohydrate intake and Betaquik tolerability. Final blood and urine samples will be taken for clinical safety assessment and routine anthropometry measurements taken.

Statistics and Plans for Analysis: This is an exploratory pilot study and its primary aim is to determine the acceptability, adherence and tolerance of the MAD with Betaquik as an adjunct therapy. A t-test and chi-square will be used with the quantitative measures, under the direction of a biostatistician. Qualitative measures will be described in a narrative summarizing the study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy; suffering from recurrent seizures (> or equal to 2 seizures per month) despite at least two anticonvulsant medication trials.
* Aged 18 years and above.
* Not on the ketogenic diet.
* Absence of any metabolic or mitochondrial disorder that precludes the use of MCT and the ketogenic diet.
* Willingly given, written, informed consent from the patient or caregiver.
* Ability to comply with study protocol and keep written records.

Exclusion Criteria:

* Non-compliant with previously recommended treatments.
* Significantly underweight (BMI <18.5), untreated dysphagia, or severe gastroesophageal reflux.
* Kidney disease, including history of nephrolithiasis.
* Uncontrolled or untreated hypercholesterolemia (>300mg/dL) or hypertriglyceridemia (>200mg/dL) within the last two years.
* Prior use of Betaquik at any time for any duration.
* Any serious medical, psychological, or social condition precluding the study intervention.
* Use of additional macro/micronutrient supplement during the study period, unless clinical indicated and prescribed by the investigator (must be recorded electronic medical records).
* Women who are pregnant/breastfeeding at the start of the study or planning to become pregnant during the study period.
* N.B.: Women who become pregnant unexpectedly during this study may, in consultation with their doctor, continue on the study's dietary product if they wish but will not have any investigations that would not normally be carried out during pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence to the MAD supplemented with Betaquik compared to previously reported historical adherence with the MAD with no MCT added. | up to 52 weeks
  Adherence will be measured by the percent of time the participant drinks Betaquik averaged over 3 months. The participant will be considered adherent if they drink the required amount on more than 80% of the prescribed days.

SECONDARY OUTCOMES:
Impact of Childhood Neurologic Disability Scale (ICNDS) | up to 52 weeks
  The Impact of Childhood Neurologic Disability Scale (ICNDS) measures factors that play a significant impact on the life of individuals with epilepsy: epilepsy, cognition, behavioral, and physical/neurologic function. Each factor has the same 11 questions applicable to the past 3 months of the individuals life which are scored 0 (not at all) to 3 (a lot). The maximum score in each factor is 33 and for the overall scale the score is 132; higher scores indicate greater impact. The Impact of Childhood Neurologic Disability Scale (ICNDS) includes a numeric scale of the child's overall quality of life ranging from 1 (poor) to 6 (excellent).
Zarit Burden Interview - Short Form | up to 52 weeks
  The Zarit Burden Interview - Short Form has 12 items which are scored as 0 (never) to 4 (nearly always). The total score ranges 0 to 48. A score for no to mild caregiver burden has a score of 0-10, mild to moderate caregiver burden a score of 10-20, and high caregiver burden a score >20.

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County + University of Southern California (LAC+USC) Medical Center, Los Angeles, California, United States